CLINICAL TRIAL: NCT03040284
Title: Non Invasive Measurements of Intracranial Pressure After Aneurysmal Subarachnoid Hemorrhage
Acronym: HEMAPIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-301; 2014-A01300-47 (Other: 2014-A01300-47)
Record Dates: First submitted 2017-01-26; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage, Familial
Keywords: noninvasive monitoring; intracranial pressure; cochlear electrophysiology; aneurysmal subarachnoid haemorrhage; cerebrovascular disorders; brain diseases
MeSH Terms: conditions — Aneurysm, Intracranial Berry, 1; Cerebrovascular Disorders; Brain Diseases

STUDY DESIGN:
Masking Description: open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- aneurysmal subarachnoid hemorrhage (Experimental)
  Interventions: Device: Echodia® hand-held equipment (ELIOS)

INTERVENTIONS:
Device: Echodia® hand-held equipment (ELIOS)

SUMMARY:
In patients at risk of increased intracranial pressure (ICP), ICP measurements require invasive transducers, usually with insertion of a catheter into the cranium, or through a spinal tap. These invasive modalities involve risks and pain and they can be done only in specialized care units, with a high associated cost.

A novel method for detecting changes in ICP has developed recently. The auditory hair cells emit sounds and electric signals in response to sound, which can be easily detected and measured non-invasively with the help of a microphone probe placed in the external ear canal or regular electrodes. Indeed, the cochlear aqueduct connects the cerebrospinal fluid (CSF) spaces to the inner ear in such a way that ICP and inner-ear fluid pressure equalize within seconds.

The evaluation of intracranial hypertension by increased ICP (invasive) is not systematically used after aneurysmal subarachnoid hemorrhage. It is then detected by using routine clinical signs of hydrocephalus or another disorder of cerebrospinal liquid flow, in combination with a standard imaging method (TDM).

The measurement of noninvasive ICP could allow earlier detection of hydrocephalus or another disorder of cerebrospinal liquid flow, and evaluate whether the increase in ICP precedes patient clinical worsening and / or imaging.

DETAILED DESCRIPTION:
In patients at risk of increased intracranial pressure (ICP), ICP measurements require invasive transducers, usually with insertion of a catheter into the cranium, or through a spinal tap. These invasive modalities involve risks and pain and they can be done only in specialized care units, with a high associated cost.

A novel method for detecting changes in ICP has developed recently. The auditory hair cells emit sounds and electric signals in response to sound, which can be easily detected and measured non-invasively with the help of a microphone probe placed in the external ear canal or regular electrodes. Indeed, the cochlear aqueduct connects the cerebrospinal fluid (CSF) spaces to the inner ear in such a way that ICP and inner-ear fluid pressure equalize within seconds.

The evaluation of intracranial hypertension by increased ICP (invasive) is not systematically used after aneurysmal subarachnoid hemorrhage. It is then detected by using routine clinical signs of hydrocephalus or another disorder of cerebrospinal liquid flow, in combination with a standard imaging method (TDM).

The measurement of noninvasive ICP could allow earlier detection of hydrocephalus or another disorder of cerebrospinal liquid flow, and evaluate whether the increase in ICP precedes patient clinical worsening and / or imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients which had recently (few days) aneurysmal subarachnoid hemorrhage
* Valid tympanometry test at least for one ear
* Between 18 and 75 years of age
* Cochlear response useful at least for an ear which has validate the tympanometry test
* Written informed consent reviewed and signed by patient
* Affiliation to a social security scheme

Exclusion Criteria:

* Invalid tympanometry test for the both ears
* Collect of cochlear responses impossible for the ear or both ear which validate the tympanometry test
* Patient refusal after enlightened information

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Presence of an intracranial pressure variation or increase | at day 1
  Presence of an intracranial pressure variation or increase when physician has diagnosed a clinical or imaging disorder of the cerebrospinal liquid flow with standard diagnose methods (composite outcome measure): clinical signs, TDM and assessment of bifrontal index.

SECONDARY OUTCOMES:
Evolution of ICP before and after the development of disorder of the cerebrospinal liquid flow according to clinical sign and/or TDM. | at day 1
Efficiency of the measurement device on repetitive measurement during one year as evaluated by composite outcome measure: clinical signs, TDM. | at day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France